CLINICAL TRIAL: NCT01483144
Title: Phase III Trial of the Safety and Efficacy of Eflornithine Combined With Sulindac Compared to Eflornithine, Sulindac as Single Agents in Patients With Familial Adenomatous Polyposis
Brief Title: Trial of Eflornithine Plus Sulindac in Patients With Familial Adenomatous Polyposis (FAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Prevention Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPP-FAP-310
Record Dates: First submitted 2011-11-21; First posted 2011-12-01 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial Adenomatous Polyposis; Eflornithine; Sulindac
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Eflornithine; Sulindac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eflornithine plus Sulindac (Experimental): Eflornithine 750 mg and Sulindac 150 mg
  Interventions: Drug: Eflornithine; Drug: Sulindac 150 MG
- Eflornithine plus Sulindac Placebo (Active Comparator): Eflornithine 750 mg and Placebo
  Interventions: Drug: Eflornithine; Drug: Sulindac placebo
- Sulindac plus Eflornithine Placebo (Active Comparator): Sulindac 150 mg and Placebo
  Interventions: Drug: Eflornithine Placebo; Drug: Sulindac 150 MG

INTERVENTIONS:
Drug: Eflornithine — Eflornithine [250 mg tablet, three tablets (750 mg) orally once a day]
  Other Names: CPP-1X
  Arms: Eflornithine plus Sulindac; Eflornithine plus Sulindac Placebo
Drug: Eflornithine Placebo — Eflornithine placebo [three tablets orally once a day]
  Other Names: CPP-1X placebo
  Arms: Sulindac plus Eflornithine Placebo
Drug: Sulindac 150 MG — Sulindac [one tablet orally once a day]
  Other Names: Clinoril
  Arms: Eflornithine plus Sulindac; Sulindac plus Eflornithine Placebo
Drug: Sulindac placebo — Sulindac placebo [one tablet orally once a day]
  Arms: Eflornithine plus Sulindac Placebo

SUMMARY:
The purpose of this randomized, double-blind, Phase III trial is to determine if the combination of eflornithine plus sulindac is superior to sulindac or eflornithine as single agents in delaying time to the first occurrence of any FAP-related event. This includes: 1) FAP related disease progression indicating the need for excisional intervention involving the colon, rectum, pouch, duodenum and/or 2) clinically important events which includes progression to more advanced duodenal polyposis, cancer or death.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of phenotypic classical FAP with disease involvement of the duodenum and/or colon/rectum/pouch.

  1. Genotype: Adenomatous polyposis coli (APC) mutation (with or without family history) required
  2. Classical FAP Phenotype: 100's to 1,000's of colorectal adenomatous polyps, usually appearing in teenage years
* Upper gastrointestinal (UGI) endoscopy/ lower gastrointestinal (LGI) endoscopy (proctoscopy/colonoscopy) performed within 30 days of randomization.
* Patients with an intact colon/rectum, except for clinical polyposis, and prophylactic surgery is being considered as a stratification site.
* Rectal/pouch polyposis as a stratification site as follows:

  1. At least three years since colectomy with ileorectal anastamosis (IRA)/proctocolectomy with pouch, and demonstrating polyposis as defined by Stage 1, 2, 3, of the proposed InSiGHT 2011 Staging System (Appendix B) and summarized as follows:

     Stage 1: 10-25 polyps, all < 5 mm Stage 2: 10-25 polyps, at least one > 1 cm Stage 3: >25 polyps amenable to complete removal, or any incompletely removed sessile polyp, or any evidence of high grade dysplasia, even if completely removed. [Note: For staging purposes only.]
  2. For all subjects, any rectal/pouch polyps > 5 mm must be excised at "baseline".
* Duodenal polyposis as a stratification site; one or more of the following:

  1. Current Spigelman Stage 3 or 4.
  2. Prior surgical endoscopic intervention within the past six months for Spigelman Stage 3 or 4 that may have been down staged to Spigelman Stage 1 or 2.
* Hematopoietic Status (within 30 days prior to randomization):

  1. No significant hematologic abnormalities
  2. White blood cell count (WBC) at least 3,000/mm3
  3. Platelet count at least 100,000/mm3
  4. Hemoglobin at least 10.0 g/dL
  5. No history of clinical coagulopathy
* Hepatic Status (within 30 days prior to randomization):

  1. Bilirubin no greater than 1.5 times ULN
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) no greater than 1.5 times ULN
  3. Alkaline phosphatase no greater than 1.5 times ULN
* Renal Status (within 30 days prior to randomization):

  a) Creatinine no greater than 1.5 times ULN
* Hearing:

  a) No clinically significant hearing loss, defined in Section 6.2, number 9.
* If female, neither pregnant nor lactating.
* Negative pregnancy test if female of child-bearing potential. Fertile patients must use effective contraception*.
* Absence of gross blood in stool; red blood on toilet paper only acceptable.
* No discrete gastric or duodenal ulcer greater than 5 mm within the past year except Helicobacter pylori-related peptic ulcer disease treated with antibiotics.
* No invasive malignancy within the past 5 years except resected non-melanomatous skin cancer, papillary thyroid cancer, or precancerous cervical dysplasia.
* No other significant medical or psychiatric problems that would preclude study participation or interfere with capacity to give informed consent.
* Use of 81-100 mg daily aspirin or up to 700 mg aspirin not more than once a week are eligible.
* No concurrent warfarin, fluconazole, lithium, Pradaxa® or other direct thrombin inhibitors, Plavix®, cyclosporine, other NSAIDs (such as ibuprofen, aspirin, diflunisal), diuretics (furosemide and thiazides), dimethylsulfoxide (DMSO), methotrexate, probenecid, propoxyphene hydrochloride, Tylenol® (acetaminophen) preparations containing aspirin or cytotoxic chemotherapy drugs.
* Willingness to forego concurrent use of supplements containing omega-3 fatty acids, corticosteroids, non-steroidal anti-inflammatory drugs or other FAP directed drug therapy.
* Able to provide informed consent and follow protocol requirements.

Exclusion Criteria:

* Prior pelvic irradiation.
* Patients receiving oral corticosteroids within 30 days of enrollment.
* Treatment with other investigational agents in the prior 4 weeks.
* Use of other non-steroidal anti-inflammatory drugs (such as ibuprofen) exceeding 4 days per month, in the prior 6 weeks.
* Regular use of aspirin in excess of 700 mg per week.
* Treatment with other FAP directed drug therapy (including sulindac or celecoxib, fish oil) within 12 weeks of study enrollment.
* Hypersensitivity to cyclooxygenase-2 inhibitors, sulfonamides, NSAIDs, or salicylates; NSAID associated symptoms of gastritis.
* Patients must not have cardiovascular disease risk factors as defined below:

  * Uncontrolled high blood pressure (systolic blood pressure > 150 mm Hg
  * Unstable angina
  * History of documented myocardial infarction or cerebrovascular accident
  * New York Heart Association Class III or IV heart failure
  * Known uncontrolled hyperlipidemia defined as LDL-C >= 190 mg/dL or triglycerides >= 500 mg/dL
* Patients with significant hearing loss are not eligible for study participation defined as hearing loss that affects everyday life and/or for which a hearing aid is required.
* Colon/rectum/pouch with high grade dysplasia or cancer on biopsy or a large polyp (>1 cm) not amenable to complete removal.
* Duodenal cancer on biopsy.
* Intra-abdominal desmoid disease, stage III or IV
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-10; Primary Completion 2018-11 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Burke, M.D., Principal Investigator — The Cleveland Clinic; James Church, M.D., Principal Investigator — The Cleveland Clinic; Gabriella Möslein, M.D., Principal Investigator — Helios Hospital
Locations (17):
- United States (10):
  - University of California San Diego, La Jolla, California
  - Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah- Huntsman Cancer Institute, Salt Lake City, Utah
- UZ Leuven, Leuven, Belgium
- Zane Cohen Centre For Digestive Diseases, Toronto, Ontario, Canada
- University Hospital Bonn, Bonn, Germany
- Academic Medical Centre, Amsterdam, Netherlands
- Institut de Malalties Digestives, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - Institute of Genetic Medicine, Newcastle upon Tyne, Tyne and Wear
  - Manchester Center for Genomic Medicine, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke CA, Dekker E, Samadder NJ, Stoffel E, Cohen A. Efficacy and safety of eflornithine (CPP-1X)/sulindac combination therapy versus each as monotherapy in patients with familial adenomatous polyposis (FAP): design and rationale of a randomized, double-blind, Phase III trial. BMC Gastroenterol. 2016 Aug 2;16(1):87. doi: 10.1186/s12876-016-0494-4. PMID 27480131
- [Result] Burke CA, Dekker E, Lynch P, Samadder NJ, Balaguer F, Huneburg R, Burn J, Castells A, Gallinger S, Lim R, Stoffel EM, Gupta S, Henderson A, Kallenberg FG, Kanth P, Roos VH, Ginsberg GG, Sinicrope FA, Strassburg CP, Van Cutsem E, Church J, Lalloo F, Willingham FF, Wise PE, Grady WM, Ford M, Weiss JM, Gryfe R, Rustgi AK, Syngal S, Cohen A. Eflornithine plus Sulindac for Prevention of Progression in Familial Adenomatous Polyposis. N Engl J Med. 2020 Sep 10;383(11):1028-1039. doi: 10.1056/NEJMoa1916063. PMID 32905675
- [Derived] Balaguer F, Stoffel EM, Burke CA, Dekker E, Samadder NJ, Van Cutsem E, Lynch PM, Wise PE, Huneburg R, Lim RM, Boytim ML, Du W, Bruckheimer EM, Cohen A, Church J; FAP-310 Investigators. Combination of Sulindac and Eflornithine Delays the Need for Lower Gastrointestinal Surgery in Patients With Familial Adenomatous Polyposis: Post Hoc Analysis of a Randomized Clinical Trial. Dis Colon Rectum. 2022 Apr 1;65(4):536-545. doi: 10.1097/DCR.0000000000002095. PMID 34261858

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo
Started | 56 | 57 | 58
Completed | 41 | 44 | 43
Not Completed | 15 | 13 | 15
Not completed — Adverse Event | 9 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 2 | 5
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 1
Not completed — Protocol Violation | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo | Total
Number analyzed (Participants) | 56 | 57 | 58 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (13.35) | 39.7 (14.76) | 38.1 (13.66) | 38.5 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 21 | 72
  Male | 34 | 28 | 37 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 3 | 13
  Not Hispanic or Latino | 50 | 50 | 54 | 154
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 3 | 10
  White | 48 | 54 | 50 | 152
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 4 | 16
  Netherlands | 4 | 6 | 5 | 15
  Belgium | 1 | 3 | 0 | 4
  United States | 31 | 30 | 42 | 103
  United Kingdom | 3 | 3 | 2 | 8
  Germany | 9 | 6 | 4 | 19
  Spain | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any FAP-related Event.
Description: Progression of disease by evaluation of FAP-related events over the course of study treatment
Time Frame: Up to 48 months from the start of treatment
Population: Intent to treat population with 171 subjects. Intent to treat population with lower GI anatomy (ower GI population) to evaluate lower GI FAP related events with 158 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo
Number analyzed (Participants) | 56 | 57 | 58
Participants
  Number with FAP-related events | 18 | 23 | 22
  Number with Lower GI FAP-related events: number analyzed (Participants) | 54 | 51 | 53
  Number with Lower GI FAP-related events | 2 | 10 | 9
Statistical Analysis 1: Comparison: Eflornithine Plus Sulindac vs Sulindac Plus Eflornithine Placebo; Intent to treat population with all FAP-related events; Test type: Superiority; p = 0.1210, stratified Cox proportional (Score) — The threshold for statistical significance is p=0.05; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.4 to 1.3] — Eflornithine plus sulindac is the numerator and sulindac plus eflornithine placebo is the denominator
Statistical Analysis 2: Comparison: Eflornithine Plus Sulindac vs Eflornithine Plus Sulindac Placebo; Intent to treat population with all FAP-related events; Test type: Superiority; p = 0.1076, stratified Cox proportional (Score) — The threshold for statistical significance is p=0.05; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.4 to 1.2] — Eflornithine plus sulindac is the numerator and eflornithine plus sulindac placebo is the denominator
Statistical Analysis 3: Comparison: Eflornithine Plus Sulindac vs Sulindac Plus Eflornithine Placebo; Lower GI population; Test type: Superiority; p = 0.0201, stratified Cox proportional (Score) — Threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 0.20, 95% CI 2-sided [0.0 to 0.8] — Eflornithine and sulindac is the numerator and sulindac and eflornithine placebo is the denominator. Reduction in relative risk for FAP-related events with the combination
Statistical Analysis 4: Comparison: Eflornithine Plus Sulindac vs Eflornithine Plus Sulindac Placebo; Lower GI population; Test type: Superiority; p = 0.0101, stratified Cox proportional (Score) — Threshold of significance was p=0.05; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0 to 0.7] — Eflornithine and sulindac is the numerator and eflornithine and sulindac placebo is the denominator

2. Secondary Outcome: Improvement in Investigator Upper GI Assessment
Description: Global assessment of change in upper GI polyp burden. These are binary outcomes derived from scores assigned by the investigator during each procedure, using a scale (-2, -1, 0, +1, +2) which corresponds, respectively, to the investigator's overall qualitative assessment of: much worse, worse, no change, improved, much improved. Summarizes the corresponding 6- and 12-month investigator change scores according to whether or not there was any positive improvement at either month 6 (compared to baseline) or at month 12 (compared to baseline or month 6), under the condition that there be no worsening at either timepoint.
Time Frame: through month 12 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo
Number analyzed (Participants) | 56 | 57 | 58
Participants
  Improved | 11 | 10 | 10
  Not Improved | 45 | 47 | 48
Statistical Analysis 1: Comparison: Eflornithine Plus Sulindac vs Sulindac Plus Eflornithine Placebo; Test type: Superiority; p = 0.8127, Mantel Haenszel — The threshold of significance was p=0.05
Statistical Analysis 2: Comparison: Eflornithine Plus Sulindac vs Eflornithine Plus Sulindac Placebo; Test type: Superiority; p = 0.8133, Mantel Haenszel — The threshold for significance was p=0.05

3. Secondary Outcome: Improvement in Investigator Lower GI Assessment
Description: Global assessment of change in lower GI polyp burden. These are binary outcomes derived from scores assigned by the investigator during each procedure, using a scale (-2, -1, 0, +1, +2) which corresponds, respectively, to the investigator's overall qualitative assessment of: much worse, worse, no change, improved, much improved. Summarizes the corresponding 6- and 12-month investigator change scores according to whether or not there was any positive improvement at either month 6 (compared to baseline) or at month 12 (compared to baseline or month 6), under the condition that there be no worsening at either timepoint.
Time Frame: through month 12 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo
Number analyzed (Participants) | 56 | 57 | 58
Participants
  Improved | 22 | 16 | 22
  Not Improved | 34 | 41 | 36
Statistical Analysis 1: Comparison: Eflornithine Plus Sulindac vs Sulindac Plus Eflornithine Placebo; Test type: Superiority; p = 0.999, Mantel Haenszel — The threshold for significance was p=0.05
Statistical Analysis 2: Comparison: Eflornithine Plus Sulindac vs Eflornithine Plus Sulindac Placebo; Test type: Superiority; p = 0.2152, Mantel Haenszel — The threshold for significance was p=0.05

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Review of adverse events monthly
Arm/Group | Eflornithine Plus Sulindac | Eflornithine Plus Sulindac Placebo | Sulindac Plus Eflornithine Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/57
Serious Adverse Events (participants affected / at risk) | 11/56 | 14/56 | 11/57
Other Adverse Events (participants affected / at risk) | 52/56 | 49/56 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eflornithine Plus Sulindac (N=56) | Eflornithine Plus Sulindac Placebo (N=56) | Sulindac Plus Eflornithine Placebo (N=57)
small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 1 (1) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
post operative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
seroma (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
abortion spontaneous (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eflornithine Plus Sulindac (N=56) | Eflornithine Plus Sulindac Placebo (N=56) | Sulindac Plus Eflornithine Placebo (N=57)
iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 4 (4)
diarrhoea (Gastrointestinal disorders) | 7 (8) | 8 (12) | 6 (9)
nausea (Gastrointestinal disorders) | 12 (18) | 9 (14) | 12 (21)
abdominal pain (Gastrointestinal disorders) | 8 (13) | 4 (4) | 8 (10)
vomiting (Gastrointestinal disorders) | 6 (8) | 7 (10) | 10 (23)
abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 4 (4) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 2 (4) | 5 (5) | 5 (6)
rectal haemorrhage (Gastrointestinal disorders) | 7 (8) | 4 (7) | 7 (8)
haematochezia (Gastrointestinal disorders) | 6 (10) | 6 (8) | 2 (3)
constipation (Gastrointestinal disorders) | 3 (4) | 5 (7) | 2 (3)
abdominal distension (Gastrointestinal disorders) | 2 (2) | 5 (6) | 3 (3)
flatulence (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (3)
pouchitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 3 (6) | 1 (1) | 2 (2)
gastritis erosive (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
fatigue (General disorders) | 4 (5) | 8 (11) | 8 (9)
influenza like illness (General disorders) | 5 (7) | 5 (7) | 3 (4)
oedema peripheral (General disorders) | 0 (0) | 3 (4) | 1 (1)
seasonal allergy (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
nasopharyngitis (Infections and infestations) | 6 (12) | 10 (14) | 4 (4)
upper respiratory tract infection (Infections and infestations) | 8 (14) | 2 (3) | 8 (10)
sinusitis (Infections and infestations) | 4 (4) | 5 (5) | 2 (3)
influenza (Infections and infestations) | 4 (4) | 3 (5) | 3 (3)
urinary tract infection (Infections and infestations) | 2 (2) | 4 (5) | 2 (2)
bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
gastroenteritis (Infections and infestations) | 7 (9) | 4 (4) | 5 (6)
gastroenteritis viral (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
weight increased (Investigations) | 2 (2) | 3 (3) | 1 (1)
platelet count decreased (Investigations) | 0 (0) | 1 (1) | 3 (4)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 5 (5)
vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 5 (6) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (8) | 3 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 2 (2)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 8 (11) | 5 (6) | 11 (12)
dizziness (Nervous system disorders) | 4 (4) | 6 (11) | 4 (6)
disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
depression (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)
anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (6)
insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 4 (4)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 2 (2)
pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 4 (4)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3)
urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT01483144/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT01483144/SAP_001.pdf